CLINICAL TRIAL: NCT03271970
Title: The Anatomic Determinants of Perforation Induced Hearing Loss
Status: Withdrawn | Type: Observational
Why Stopped: PI no longer wishes to conduct the study. No participants were enrolled.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00073436
Record Dates: First submitted 2017-08-17; First posted 2017-09-05 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2018-01

CONDITIONS: Conductive Hearing Loss; Perforated Tympanic Membrane
MeSH Terms: conditions — Hearing Loss, Conductive; Tympanic Membrane Perforation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with conductive hearing loss

SUMMARY:
The purpose of this study is to identify factors that may contribute to conductive hearing loss. Conductive hearing loss is a type that is due to a problem with the outer or middle ear. Because of this, sound does not travel through the ear normally. Perforated tympanic membranes of study patients will be photographed during the patient's routine visit using a digital otoscope. These pictures will be used to analyze perforation size as an absolute value as well as a percentage of the tympanic membrane. Audiometric results and CT scans of temporal bone (reports and images) collected as standard of care will be evaluated. Images of CT scans will be imported into a medical imaging software for creation of anatomically realistic 3D models of the middle ear and mastoid air space. Structural analysis on each 3D model will be conducted and analyzed, the volume of middle ear and mastoid air spaces will be recorded, and data points will be correlated with perforation size and location to audiogram results.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 89 years of age
* Confirmed diagnosis of conductive hearing loss secondary to tympanic membrane perforation
* Treated for the above condition by a Duke physician
* Received both a CT temporal bone scan interpreted by a Duke radiologist and audiometry at a Duke-based facility (both tests performed within four weeks of each other), as part of standard pre-operative workup

Exclusion Criteria:

* Temporal CT scan with inadequate resolution as per determination of study staff
* Unable to provide written informed consent
* Unable to read and understand English

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with conductive hearing loss due to tympanic membrane perforation.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-04 (Estimated); Primary Completion 2018-01-03 (Actual); Study Completion 2018-01-03 (Actual)

PRIMARY OUTCOMES:
presence of perforation | Day 1
  Number of patients with perforations
absence of perforation | Day 1
  number of patients without perforations
change in audiometric measurements | Baseline, up to 16 weeks
  looking at difference between baseline and last observation

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Frank-Ito, PhD, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No